CLINICAL TRIAL: NCT00596778
Title: Chest Physiotherapy on Immediate Postoperative in Patients Submitted to High Abdominal Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: terminated
Sponsor: University of Sao Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Roberta Munhoz Manzano, Chest physiotherapy on immediate postoperative in patients submitted to high abdominal surgery, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPPesq836/03; CAPPesq836/03
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2008-01

CONDITIONS: Abdominal Surgery; Spirometry; Chest Physiotherapy
Keywords: Physical therapy specialty; Postoperative period. Abdominal surgery; Anesthesia recovery period; Spirometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- C, CP (Other): Thirty-one adults were randomly assigned to control (C) and chest physiotherapy (CP) groups. Chest physiotherapy group received treatment at the post-anesthesia unit care and control group did not.
  Interventions: Other: chest physiotherapy

INTERVENTIONS:
Other: chest physiotherapy — The protocol consisted of breathing exercises during 30 minutes and included: passive and localized exercises, deep diaphragmatic breathing and exercises of chest wall expansion.

SUMMARY:
Abdominal surgical procedures can increase risks of pulmonary complications.The aim of the study was to evaluate the benefits of an early intervention of chest physiotherapy during immediate post-operative in patients submitted to elective abdominal surgery.

DETAILED DESCRIPTION:
Thirty-one adults were randomly assigned to control and chest physiotherapy groups. Spirometry, pulse oximetry and anamneses were performed before (pre-operative) and in the second post-operative day. Chest physiotherapy group received treatment at the post-anesthesia unit care and control group did not. Chest physiotherapy improved oxygen-hemoglobin saturation in elective post-operative abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Pre-operative for elective upper abdominal surgery, such as - hernia repair, gall bladder or large bowel removal, exploratory laparotomy, and submitted to general anesthesia or other interventions in abdominal cavity accomplished by conventional laparotomy

Exclusion Criteria:

* Patients with indication of liver transplant or bearers of aneurysm of any arterial segment.
* Patients submitted to video-laparoscopy surgery.

Ages: 21 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2004-02; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Effective of chest physiotherapy before and after surgery | 3 days (before surgery - second post operative)